CLINICAL TRIAL: NCT00115869
Title: Hutchinson Smoking Prevention Project
Acronym: HSPP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Arthur V. Peterson, Jr., PhD, Fred Hutchinson Cancer Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FHCRC IRB #324; R01CA038269 (NIH)
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Results first posted 2012-11-29 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-10

CONDITIONS: Smoking Among Youth
Keywords: smoking prevention; tobacco use prevention; adolescent tobacco use; prevention intervention
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No-intervention control (No Intervention)
- Social influences school-based smoking prevention curriculum (Experimental)
  Interventions: Behavioral: Social-influences

INTERVENTIONS:
Behavioral: Social-influences — grades 3-10, school-based social influences tobacco use prevention curriculum
  Arms: Social influences school-based smoking prevention curriculum

SUMMARY:
The Hutchinson Smoking Prevention Project is a 16-year, group-randomized trial to determine the extent to which a school-based (grades 3-10), theory-based, social-influences tobacco use prevention intervention can deter youth tobacco use throughout and beyond high school.

DETAILED DESCRIPTION:
Cigarette smoking remains the number one cause of preventable premature death in the U.S., annually killing more than 400,000 Americans. Without reversal of adolescent smoking trends, five million of today's youth will die prematurely of smoking-related illnesses. The 16-year Hutchinson Smoking Prevention Project (HSPP) was conducted in 1984-1999 to (1) address challenges of trial design and execution in school-based smoking prevention by developing the most rigorous school-based randomized trial possible, and (2) use the trial to answer the scientific questions, "To what extent can a theory-based, social-influences smoking prevention intervention spanning elementary, middle and high school grades reduce smoking among youth at 12th grade and two years post-high-school?"

The HSPP trial used a group-randomized, matched pair design with the school district as the experimental unit. Of 40 participating school districts, 20 were randomly assigned to the experimental (intervention) condition and 20 were assigned to the control (no HSPP intervention) condition. No restrictions were placed on the health promotion or tobacco use prevention activities of the control districts, thus enabling schools to continue whatever health curricula were normally offered. Main endpoints were daily smoking at 12th grade and 2 years after high school (Plus-2). Study participants (N=8,388) were two consecutive third grade enrollments in each of the 40 school districts. All third graders were followed to endpoint, including those who dropped out of school or otherwise left their school districts. The study achieved a 94% follow-up rate at the Plus-2 endpoint.

The HSPP intervention was a teacher-led, grades 3-10 tobacco use prevention curriculum plus unit-specific teacher training. There were 65 classroom lessons in the HSPP curriculum: 9 lessons in each of grades 3-5, 10 lessons in each of grades 6-7, 8 lessons in grade 8, and 5 lessons in each of grades 9-10, for a total number of 46.75 hours of classroom instruction time in grades 3-10. The HSPP uses an enhanced social influences approach that includes the 15 NCI-endorsed "essential elements" for school-based tobacco prevention and meets the CDC's "best practices" guidelines. The intervention's behavioral components featured skills for identifying and resisting social influences to smoke, correcting erroneous normative perceptions regarding smoking, promoting tobacco-free norms, and building self-efficacy for tobacco-free lifestyle choices. The intervention was developed to be practical for the school setting, emphasizing ease of use by teachers, good fit into school routines and with schools' existing educational objectives, and incorporation of topics/activities that are interesting, engaging and developmentally-appropriate for students.

ELIGIBILITY:
Inclusion Criteria:

* All students enrolled in third grade in one of two consecutive classes of third graders in an HSPP participating Washington school district (1984-85; 1985-86; 1986-87).

Exclusion Criteria:

* Enrolled but classified by participating school district as developmentally unable to learn.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8388 (Actual)
Dates: Start 1984-09; Primary Completion 1999-08 (Actual); Study Completion 1999-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur V. Peterson, Jr., PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Background] Peterson AV, Mann SL, Kealey KA, Marek PM. Experimental design and methods for school-based randomized trials. Experience from the Hutchinson Smoking Prevention Project (HSPP). Control Clin Trials. 2000 Apr;21(2):144-65. doi: 10.1016/s0197-2456(99)00050-1. PMID 10715512
- [Background] Kealey KA, Peterson AV Jr, Gaul MA, Dinh KT. Teacher training as a behavior change process: principles and results from a longitudinal study. Health Educ Behav. 2000 Feb;27(1):64-81. doi: 10.1177/109019810002700107. PMID 10709793
- [Background] Burt RD, Dinh KT, Peterson AV Jr, Sarason IG. Predicting adolescent smoking: a prospective study of personality variables. Prev Med. 2000 Feb;30(2):115-25. doi: 10.1006/pmed.1999.0605. PMID 10656839
- [Background] Mann SL, Peterson AV Jr, Marek PM, Kealey KA. The Hutchinson Smoking Prevention Project trial: design and baseline characteristics. Prev Med. 2000 Jun;30(6):485-95. doi: 10.1006/pmed.2000.0664. PMID 10901491
- [Background] Burt RD, Peterson AV Jr. Smoking cessation among high school seniors. Prev Med. 1998 May-Jun;27(3):319-27. doi: 10.1006/pmed.1998.0269. PMID 9612822
- [Result] Peterson AV Jr, Kealey KA, Mann SL, Marek PM, Sarason IG. Hutchinson Smoking Prevention Project: long-term randomized trial in school-based tobacco use prevention--results on smoking. J Natl Cancer Inst. 2000 Dec 20;92(24):1979-91. doi: 10.1093/jnci/92.24.1979. PMID 11121460
- See also: Web site of the Fred Hutchinson Cancer Research Center — http://www.fhcrc.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited as 3rd graders in the consecutive years from 40 collaborating school districts in Washington State. The study participants were recruited in 3 waves: Wave I, 6 school districts (1984 and 1985); Wave II, 14 school districts (1985 and 1986); and Wave III, 20 school districts (1986 and 1987).
Pre-assignment Details: Forty-two (42) children were not eligible for the study because they were considered by their schools to be developmentally unable to learn.
Groups:
- No-intervention Control: No-intervention control group
- Grade 3-12 School-based Intervention: Grade 3-12 school-influences school-based smoking prevention intervention
Period: Overall Study
Arm/Group | No-intervention Control | Grade 3-12 School-based Intervention
Started | 4211 | 4177
Completed Data Collection at 12th Grade | 3876 | 3847
Completed | 3894 | 3881 (Follow-up at two years post high school.)
Not Completed | 317 | 296

BASELINE CHARACTERISTICS:
Groups:
- Social Influences School-based Smoking Prevention Curriculum: Social influences school-based smoking prevention curriculum group
- Total: Total of all reporting groups
Arm/Group | No-intervention Control | Social Influences School-based Smoking Prevention Curriculum | Total
Number analyzed (Participants) | 4211 | 4177 | 8388
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4211 | 4177 | 8388
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2058 | 2073 | 4131
  Male | 2153 | 2104 | 4257
Region of Enrollment [Number; unit: participants]
  United States | 4211 | 4177 | 8388

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Smoking Daily at 12th Grade
Description: Response "1 to 3 cigarettes per day," "4 to 10 cigarettes per day," "11 to 20 cigarettes per day," or "More than 20 cigarettes per day" to the Item "How often do you currently smoke cigarettes?"
Time Frame: 12th grade
Measure: Number; unit: participants
Groups:
- No-intervention Control: No-intervention control condition
- Social Influences School-based Smoking Prevention Curriculum: School-based social-influences smoking prevention curriculum condition
Arm/Group | No-intervention Control | Social Influences School-based Smoking Prevention Curriculum
Number analyzed (Participants) | 3876 | 3847
participants | 995 | 976

2. Primary Outcome: Whether or Not Smoking Daily at 2 Years After High School
Description: Response (from the 2-years-after-high school questionnaire) "Daily: 1 to 10 cigarettes a day," "Daily: 11 to 20 cigarettes a day," "Daily: more than a pack a day" to the Item "How often do you currently smoke cigarettes?"
Time Frame: 2 years after high school
Measure: Number; unit: participants
Groups:
- School-based Smoking Prevention Curriculum: Social influences school-based smoking prevention curriculum group
Arm/Group | No-intervention Control | School-based Smoking Prevention Curriculum
Number analyzed (Participants) | 3894 | 3881
participants | 1132 | 1103

ADVERSE EVENTS:
Groups:
- No-intervention Control Group: no-intervention control
- School-based Smoking Prevention Curriculum Group: school-based smoking prevention curriculum
Arm/Group | No-intervention Control Group | School-based Smoking Prevention Curriculum Group
Serious Adverse Events (participants affected / at risk) | 0/4211 | 0/4177
Other Adverse Events (participants affected / at risk) | 0/4211 | 0/4177

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No